CLINICAL TRIAL: NCT02017938
Title: Establishing the Central and Peripheral Fatigue Indexes and VR Based Anti-fatigue Training Paradigm for Individuals With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Profesor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101-5141B
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Parkinson's Disease (PD)
Keywords: Fatigue; electromyography (EMG); central fatigue; cycling training
MeSH Terms: conditions — Parkinson Disease; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Stage 1: Health group (No Intervention): To establish non-invasive fatigue monitoring method via testing healthy individuals.
- Stage 2: PD group (Experimental): To find the optimal feedback variables for anti-fatigue training on individuals with PD.
  Interventions: Procedure: Virtual Reality anti-fatigue ergo cycling training (Self-made)
- Stage 2: Health group (Experimental): Stage 2 controlled group
  Interventions: Procedure: Virtual Reality anti-fatigue ergo cycling training (Self-made)
- Stage 3: PD group (Experimental): To evaluate the effect of four weeks of VR anti-fatigue ergo cycling training on various fatigue components and functional abilities in individuals with PD.
  Interventions: Procedure: Virtual Reality anti-fatigue ergo cycling training (Self-made)
- Stage 3: PD controlled group (No Intervention): Stage 3 controlled group

INTERVENTIONS:
Procedure: Virtual Reality anti-fatigue ergo cycling training (Self-made) — To establish a Virtual Reality systems to reduce fatigue of cycling training for PD subjects.
  Arms: Stage 2: Health group; Stage 2: PD group; Stage 3: PD group

SUMMARY:
Fatigue is one of the most common symptoms in individuals with Parkinson's Disease (PD). Past researches indicated that more than half of the individuals with PD demonstrated fatigue symptom. The severity of fatigue was also correlated to the quality of life in individuals with PD. Finding the contributions of the central and the peripheral factors to fatigue, building reliable fatigue indexes, and developing an effective training program for individuals with PD are very important.

The purpose of this project is to develop non-invasive method to monitor central and peripheral fatigue, to establish Virtual Reality(VR) anti-fatigue ergo cycling training paradigm, and to evaluate the long term training effect in individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson disease
* Hoehn and Yahr ≦3

Exclusion Criteria:

* Musculoskeletal injuries
* Osteoporosis
* Diabetes
* Any peripheral or central nervous system injury or disease patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-12-10 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Muscle twitch force | baseline, 1 week
  Measure of changes in muscle twitch force by interpolation twitch technique.
Muscle voluntary activity level | Baseline,1 week
  Measure of changes in muscle voluntary activity level by interpolation twitch technique.
Heart rate/Heart rate variability | Baseline,1 week
  Measure of changes in Heart rate/Heart rate variability.
Borg's rate of perceived exertion | Baseline,1 week
  Measure of changes in Borg's rate of perceived exertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886